CLINICAL TRIAL: NCT02711449
Title: Preoperative Methylprednisolone to Patients Suspected of Appendicitis Undergoing Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jakob Kleif (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jakob Kleif, MD, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-810; 2015-004800-46 (EudraCT Number)
Record Dates: First submitted 2016-02-23; First posted 2016-03-17 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Suspected Appendicitis
Keywords: acute surgery; laparoscopy
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Experimental): 125 mg Methylprednisolone intravenously approximately 30 minutes prior to skin incision
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): 0.9% Saline intravenously approximately 30 minutes prior to skin incision
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Methylprednisolone — 125 mg methylprednisolone as an intravenously bolus injection approximately 30 minutes prior to skin incision.
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: 0.9% Saline — 0,9% Saline as an intravenously bolus injection approximately 30 minutes prior to skin incision.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To test whether 125 mg preoperative methylprednisolone intravenously can reduce postoperative pain after laparoscopy for suspected appendicitis and to test whether preoperative methylprednisolone can reduce postoperative fatigue, increase quality of sleep, reduce nausea or vomiting, reduce duration of convalescence and increase overall quality of recovery after laparoscopy for suspected appendicitis.

DETAILED DESCRIPTION:
Patients enrolled are randomized to active substance or placebo approximately 30 minutes prior to skin incision.

Patients are followed for 30 days postoperative with registration of outcomes on a postoperative questionnaire. Patients are contacted by telephone at every registration time. The primary outcome is also secured over the telephone in case patients do not return their questionnaire.

With a power of 80% and a significance level of 5% we need 64 patients (32 in each arm) to show a 30% reduction in postoperative pain during the first 3 postoperative days with 5 measurements and we need 42 patients (21 in each arm) to show a 15% increase in the QoR-15 during the first 3 postoperative days. With an anticipated loss to follow up of 20% we need 80 patients ( 40 in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopy for suspected appendicitis
* Age 18 years or older
* American Society of Anesthesiologist (ASA) class I-III.
* Gives written and oral consent

Exclusion Criteria:

* Known inflammatory bowel disease.
* Known autoimmune disease.
* Chronic pain patient.
* Presumed poor compliance.
* Pregnant or breastfeeding.
* In systematic treatment with glucocorticoids or other immunosuppressive treatment.
* Known renal disease, GFR<30.
* Known liver cirrhosis.
* Known heart failure, EF<40%.
* Known glaucoma.
* Known ocular herpes simplex.
* Known cushings disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pain at rest during the first 3 postoperative days on a 11-point NRS | 6 hours, 12 hours, postoperative day (POD) 1, POD2 and POD3
  Powered to detect 30% reduction, Random regression model (mixed effects model)

SECONDARY OUTCOMES:
Pain when coughing during the first 3 postoperative days on a 11-point NRS | 6 hours, 12 hours, postoperative day (POD) 1, POD2 and POD3
  Random regression model (mixed effects model)
Fatigue during the first 3 postoperative days on a 11-point NRS | 6 hours, 12 hours, postoperative day (POD) 1, POD2 and POD3
  Random regression model (mixed effects model)
Sleep during the first 3 postoperative days on a 11-point NRS | postoperative day (POD) 1, POD2 and POD3
QoR-15 during the first 3 postoperative days | postoperative day (POD) 1, POD2 and POD3
  Powered to detect 15% increase,
Incidence of postoperative nausea or vomiting during the first postoperative day | 6 hours, 12 hours and 24-32 hours postoperative
Pain at rest after POD3 on a 11-point NRS | postoperative day (POD) 7, POD 14 and POD 30
Pain when coughing after POD3 on a 11-point NRS | postoperative day (POD) 7, POD 14 and POD 30
Fatigue after POD3 on a 11-point NRS | postoperative day (POD) 7, POD 14 and POD 30
Sleep after POD3 on a 11-point NRS | postoperative day (POD) 7, POD 14 and POD 30
QoR-15 after POD 3 | postoperative day (POD) 7, POD 14 and POD 30
Mobilization during the first postoperative day on a 4-point likert scale | 6 hours, 12 hours and postoperative day 1
Resumption of occupational activity | Up to 60 days postoperative
  Number of days from surgery until resumption of occupational activities
Resumption of recreational activity | Up to 60 days postoperative
  Number of days from surgery until resumption of recreational activities
Duration of convalescence | Up to 60 days postoperative
  Number of days from surgery until resumption of both occupational and recreational activities
Adverse events according to GCP guidelines | 30 day postoperative
Postoperative complications according to the Clavien-Dindo classification | 30 day postoperative
Opioid consumption during the first 24 hours postoperative | 24 hours postoperative
  Both as a the need for opioids and the amount equivalent to intravenous morphine.
Need for rescue antiemetics during the first 24 hours postoperative | 24 hours postoperative
Duration of postoperative hospital stay | 30 days postoperative
  The duration of the postoperative hospital stay in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Kleif, M.D., Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - Nordsjaellands Hospital, Hillerød
  - Køge Sygehus, Køge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kleif J, Gogenur I. Severity classification of the quality of recovery-15 score-An observational study. J Surg Res. 2018 May;225:101-107. doi: 10.1016/j.jss.2017.12.040. Epub 2018 Feb 21. PMID 29605019
- [Derived] Kleif J, Hauge CI, Vilandt J, Gogenur I. Randomized Clinical Trial of Preoperative High-Dose Methylprednisolone on Postoperative Pain at Rest After Laparoscopic Appendectomy. Anesth Analg. 2018 May;126(5):1712-1720. doi: 10.1213/ANE.0000000000002693. PMID 29200067